CLINICAL TRIAL: NCT06977555
Title: Communication With Mechanically Ventilated Intensive Care Patients
Acronym: COMMEC-ICU
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Lovisenberg Diaconal University College (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Researcher, professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 639899
Record Dates: First submitted 2024-08-23; First posted 2025-05-18 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Communication; Intensive Care Unit Syndrome
Keywords: mechanically ventilated patients; delir; symptoms; self-efficacy
MeSH Terms: conditions — Critical Illness; Communication

STUDY DESIGN:
Intervention Model Description: We will enroll a communication intervention in five ICUs at two University Hospitals in Norway
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICU patients (No Intervention): Data on patients admitted to the ICUs will be collected before and after the intervention (the teaching program for the nurses). Two different patient samples.
- ICU nurses (Active Comparator): Data from the nurses before and after they have received the training in communication will be collected. We will include the same sample pre- and post.
  Interventions: Behavioral: Communication Course and skills training

INTERVENTIONS:
Behavioral: Communication Course and skills training — A multi module intervention where the nurses will learn about communication with mechanically ventilated patients will be developed. The investigators hypothesize that this intervention will:
  1. make it easier for mechanically ventilated ICU patients to communicate their needs and symptoms during mechanical ventilation and to improve their symptom burden.
  2. improve ICU nurses' skills in communicating with ICU patients who are unable to speak. This will potentially contribute to better communication with critically ill patients, including those being delirious.
  3. improve ICU nurses´ satisfaction with their communication.
  Arms: ICU nurses

SUMMARY:
The overarching aim of this multicenter study is to develop a multimodule training intervention (COMMEC-ICU) for nurses working in ICUs, to increase nurses skills and knowledge and then improve communication for mechanically ventilated ICU patients. The intervention will be implemented at the included ICUs and evaluated both on nurses in the ICU and patients. Patients with delirium will also be included.

DETAILED DESCRIPTION:
The specific objectives of the research proposal are to:

1. Investigate ICU patients' perceptions of communication difficulties during mechanical ventilation, and evaluate the relationship between communication difficulties and symptom burden.
2. Describe ICU nurses' communication skills, communication techniques commonly used, and satisfaction with communication with patients.

   The results from objectives 1 and 2 are of relevance as such, but will also be used as a basis to develop the COMMEC-ICU and as a pre-intervention measure prior to implementation of the new program.
3. Further develop and implement COMMEC-ICU in the selected ICUs.
4. Evaluate the effect of COMMEC-ICU on a) ICU nurses after receiving the training program b) former ICU patients that have been treated in the ICUs with were the intervention have been implemented.

ELIGIBILITY:
Inclusion Criteria patients:

* Patients over the age of 18
* First ICU admission during the hospital stay
* Cognitively competent at the time of consenting to participate
* Invasive mechanical ventilation via endotracheal tube or tracheostomy for over 48 hours or more calendar days
* Patients must have been reported awake and communicative or with a Richmond Agitation and Sedation scale over - 1.

Exclusion Criteria patients:

* Patients who cannot understand Norwegian
* Patients without an address
* Patients who have cognitive disabilities and are not able to consent or receive information about the study

Inclusion criteria nurses: having clinical experience from the ICU for more than a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Ease of Communication Scale- patients | 6-8 months before and 4 weeks after the intervention were nurses go through a training program
  10-item instrument using a 5-point Likert scale to assess communication difficulty (0 "not hard at all"; 1 "a little hard"; 2 "somewhat hard", 3 "quite hard", and 4 "extremely hard").
Nurses communication skills and satisfaction | 6-8 months before and 3 months after the intervention (communication training program)
  The scale is developed based on previous studies about communication with ICU patients. It consists of items covering self-perceived competency and satisfaction of communication skills. The scale consists of 16 questions about their satisfaction with communication on a 5 point Likert scale from "never" to "always", and 7 questions about their use of communication aids on a 5 point Likert scale from "never" to "always". The last seven items also have one option to tick "not available".

SECONDARY OUTCOMES:
10 Symptom checklist- patients | Symptom assessement will be conducted at ICU discharge, 3-6 months before and one to two months after the intervention is given to the nurses.after the intervention.
  The scale consists of 10 items, but we will only use 5 symptoms in the present study. Patients can rate whether the symptom (pain, tiredness shortness of breath, anxiety, thirst) is present (tick if yes). If present they are asled about intensity (0=not at all and 10= Very serious) and level of distress (1=not very distressing to 10=very distressing).
Symptom communication nurses | 6-8 months before the intervention and 3 months after the intervention (communication training program).
  10 questions about the communication symptoms, on a 10 point scale from extremely difficult to very easy
Norwegian version of Self-efficacy questionnaire SE-12- nurses | 6-8 months before and 3 months after the intervention (communication training program)
  The scale consists of 16 questions about self perceived competency of communication skills. The scale will be answered on a 10 point Likert scale from "not sure at all" to "very sure". Some questions about the effect of the communication and perceived use of the communication course will be added to the measurement 3 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — OUS
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SE-12 questionnaire nurses — https://bmcmededuc.biomedcentral.com/articles/10.1186/s12909-016-0798-7
- See also: 10 symptom check-list patients in the ICU — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3377582/